CLINICAL TRIAL: NCT02325739
Title: A Phase I/II, Multicenter, Open-label Study of Oral FGF401 in Adult Patients With Hepatocellular Carcinoma or Solid Malignancies Characterized by Positive FGFR4 and KLB Expression
Brief Title: FGF401 in HCC and Solid Tumors Characterized by Positive FGFR4 and KLB Expression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFGF401X2101; 2014-002929-35 (EudraCT Number)
Record Dates: First submitted 2014-12-09; First posted 2014-12-25 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma (HCC); Solid Malignancies
Keywords: FGF401; PDR001; PD-1; FGFR4; FGF19; HCC; solid malignancies characterized by positive FGFR4 and KLB expression
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — roblitinib; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Phase I: FGF401 50 mg fasted (Experimental): Participants received single agent FGF401 50 mg while fasted
  Interventions: Drug: FGF401
- Phase I: FGF401 80 mg fasted (Experimental): Participants received single agent FGF401 80 mg while fasted
  Interventions: Drug: FGF401
- Phase I: FGF401 80 mg fed (Experimental): Participants received single agent FGF401 80 mg while fed
  Interventions: Drug: FGF401
- Phase I: FGF401 120 mg fasted (Experimental): Participants received single agent FGF401 120 mg while fasted
  Interventions: Drug: FGF401
- Phase I: FGF401 120 mg fed (Experimental): Participants received single agent FGF401 120 mg while fed
  Interventions: Drug: FGF401
- Phase I: FGF401 150 mg fasted (Experimental): Participants received single agent FGF401 150 mg while fasted
  Interventions: Drug: FGF401
- Phase I: FGF401 80 mg + PDR001 300 mg (Experimental): Participants received FGF401 80 mg in combination with PDR001 300 mg while fasted
  Interventions: Drug: FGF401; Biological: PDR001
- Phase I: FGF401 120 mg + PDR001 300 mg (Experimental): Participants received FGF401 120 mg in combination with PDR001 300 mg while fasted
  Interventions: Drug: FGF401; Biological: PDR001
- Phase II: Group 1 - FGF401 120 mg QD (Experimental): Group 1 was comprised of HCC participants from Asian countries who received single agent FGF401 120 mg QD while fasted
  Interventions: Drug: FGF401
- Phase II: Group 2 - FGF401 120 mg QD (Experimental): Group 2 was comprised of HCC participants from non-Asian countries who took single agent FGF401 120 mg QD while fasted
  Interventions: Drug: FGF401
- Phase II: Group 3 - FGF401 120 mg QD (Experimental): Group 3 was comprised of participants with other solid malignancies regardless of geography who took single agent FGF401 120 mg QD while fasted
  Interventions: Drug: FGF401

INTERVENTIONS:
Drug: FGF401 — FGF401 is a FGFR4 inhibitor.
Biological: PDR001 — PDR001 is a humanized anti-PD1 IgG4 antibody that blocks the binding of PD-L1 and PD-L2
  Arms: Phase I: FGF401 120 mg + PDR001 300 mg; Phase I: FGF401 80 mg + PDR001 300 mg

SUMMARY:
Estimate the maximum tolerated dose and/or recommended phase II dose and efficacy of FGF401 as single agent and in combination with PDR001 in patients with hepatocellular carcinoma and as single agent in patients with other solid malignancies based on RECIST 1.1.

DETAILED DESCRIPTION:
The primary objectives of this study were in 2 parts: Phase l & Phase II.

The study included different periods starting by molecular pre-screening (applicable for all subjects enrolled under protocol versions 00 to 03, or applicable only for Phase I and Group 3 in Phase II of FGF401 single agent, for subjects enrolled under protocol version 04), Screening, Treatment, End of Treatment, Disease progression follow-up (if applicable), Safety follow-up and then ended by survival follow-up period

In the Phase I part, subjects with HCC or other advanced solid tumors characterized by positive FGFR4 and KLB expression were enrolled and treated with FGF401 as a single agent or in combination with PDR001. Subjects in this phase were dosed under fasted or fed conditions.

In the Phase 2 part, subjects with advanced HCC or other solid tumors bearing positive FGFR4 and KLB expression were enrolled into three groups (Group 1: HCC subjects from Asian countries; Group 2: HCC subjects from non-Asian countries; Group 3: Subjects with other solid malignancies regardless of geography) to assess the preliminary anti-tumor activity of FGF401 in Phase ll. This Phase II part investigated the anti-tumor activity of FGF401 single agent and in combination with PDR001.

Each group within the Phase II dose expansion part targeted a different number of subjects. Group 1 and Group 2 planned to enroll around 40 subjects each and Group 3 planned to enroll approximately 20 subjects. Subjects in this phase were dosed under fasted conditions.

Oral FGF401 was administered on a continuous once daily (QD) dosing regimen for both FGF401 single agent and in combination with PDR001 parts. Intravenous PDR001 was administered in a fixed dosing regimen of 300 mg iv every three weeks as per protocol until subject experienced unacceptable toxicity, progressive disease and/or treatment was discontinued at the discretion of the Investigator or withdrawal of consent.

Because the enrollment of new subjects in this study was halted for business reason on 03-Jul-2018 early enrollment termination was declared following the initial halt of enrollment once the global last subject last visit was achieved as per protocol, and consequently the phase II part of the FGF401+PDR001 combination did not start, none of the planned analyses related to the phase II part of the FGF401+PDR001 combination arm were performed.

Duration of treatment: Subjects could continue study treatment until they experienced any of the following: Disease progression (radiologically documented according to RECIST v1.1) as assessed by the Investigator, unacceptable toxicity, & treatment was discontinued at the discretion of the Investigator or the subject.

Subjects who permanently discontinued the study treatment for any reason other than disease progression or withdrawal of consent had to continue efficacy assessments as scheduled in the protocol until the time of disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG Performance Status ≤ 1
2. Presence of at least one measurable lesion according to RECIST v1.1. c-i) FGF401 single agent-Phase I and Phase II, Group 3: Patients with HCC or advanced solid tumors, who have progressed despite standard therapy or are intolerant of standard therapy, or for whom no standard therapy exists. c-ii) FGF401 single agent-Phase II, Groups 1 and 2: HCC patients previously treated with sorafenib for advanced HCC with documented disease progression during or after discontinuation of sorafenib treatment, or intolerance to sorafenib treatment c-iii) FGF401 in combination with PDR001:Advanced HCC patients who have received up to 2 previous lines of systemic treatment and one treatment must have included sorafenib with documented disease progression during or after discontinuation of sorafenib treatment, or intolerance to sorafenib treatment

Exclusion Criteria:

1. Previous treatment with a selective FGF19-FGFR4 targeted therapy and/or pan-FGFR inhibitor.
2. Symptomatic CNS metastases which are neurologically unstable or requiring increasing doses of steroids to control their CNS disease.
3. Patient having out of range laboratory values defined as:

   * Hematology Hemoglobin ≤ 9 g/dL (SI Units: 90 g/L) Platelet count < 75000/mm3 Absolute neutrophil count (ANC) < 1500/mm3
   * Chemistry Total bilirubin ≥ 2 mg/dL AST and/or ALT > 3 x ULN Serum creatinine > 1.5 x ULN and/or creatinine clearance ≤ 45 mL/min
   * Coagulation: PT > 4 seconds more than ULN or INR > 1.7
4. Pregnant or nursing (lactating) women.

Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-12-29 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (3):
  - University of California LA Santa Monica Location, Los Angeles, California
  - Massachusetts General Hospital Oncology Dept, Boston, Massachusetts
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
- Novartis Investigative Site, Shanghai, Shanghai Municipality, China
- France (5):
  - Novartis Investigative Site, Rennes, Ille Et Vilaine
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Toulouse
- Germany (4):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Japan (2):
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Chan SL, Schuler M, Kang YK, Yen CJ, Edeline J, Choo SP, Lin CC, Okusaka T, Weiss KH, Macarulla T, Cattan S, Blanc JF, Lee KH, Maur M, Pant S, Kudo M, Assenat E, Zhu AX, Yau T, Lim HY, Bruix J, Geier A, Guillen-Ponce C, Fasolo A, Finn RS, Fan J, Vogel A, Qin S, Riester M, Katsanou V, Chaudhari M, Kakizume T, Gu Y, Porta DG, Myers A, Delord JP. A first-in-human phase 1/2 study of FGF401 and combination of FGF401 with spartalizumab in patients with hepatocellular carcinoma or biomarker-selected solid tumors. J Exp Clin Cancer Res. 2022 Jun 2;41(1):189. doi: 10.1186/s13046-022-02383-5. PMID 35655320
- [Derived] Castanon Alvarez E, Giallombardo M, Gil-Bazo I, Papadimitriou K, Pauwels P, Peeters M, Rolfo C. Looking into the "Garden of the Hesperides": new drugs for hepatocellular carcinoma. Minerva Chir. 2015 Apr;70(2):119-29. Epub 2015 Jan 23. PMID 25614940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 160 subjects were enrolled & treated with FGF401 single agent. In the Phase I part 74 subjects & 86 subjects in the Phase II part. 12 subjects were treated in the Phase I of the combination of FGF401 and PDR001. All subjects completed the study as per protocol & reasons for discontinuation of treatment are provided in the 'Not Completed' section.
Pre-assignment Details: At least 21 evaluable subjects were to be treated in Phase I for the model to have reasonable operating characteristics relating to its MTD &/or RP2D. Each group in the Phase II dose expansion targeted a different number of subjects. Group 1 & Group 2 planned to enroll around 40 subjects each & Group 3 planned to enroll approximately 20 subjects.
Groups:
- Phase I: 50 mg Fasted: Participants received single agent FGF401 50 mg while fasted
- Phase I: 80 mg Fasted: Participants received single agent FGF401 80 mg while fasted
- Phase I: 80 mg Fed: Participants received single agent FGF401 80 mg while fed
- Phase I: 120 mg Fasted: Participants received single agent FGF401 120 mg while fasted
- Phase I: 120 mg Fed: Participants received single agent FGF401 120 mg while fed
- Phase I: 150 mg Fasted: Participants received single agent FGF401 150 mg while fasted
- Phase II: Group 1 - FGF401 120 mg QD: Group 1 was comprised of HCC participants from Asian contrives who took single agent FGF401 120 mg QD while fasted
- PhaseII: Group 3 - FGF401 120 mg QD: Group 3 was comprised of participants with other solid malignancies regardless of geography who took single agent FGF401 120 mg QD while fasted
Period: Phase I Part
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted | Phase I: FGF401 80 mg + PDR001 300 mg | Phase I: FGF401 120 mg + PDR001 300 mg | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD | PhaseII: Group 3 - FGF401 120 mg QD
Started | 11 | 6 | 5 | 26 | 19 | 7 | 6 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 6 | 5 | 26 | 19 | 7 | 6 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 2 | 3 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Progressive disease | 9 | 6 | 3 | 23 | 14 | 6 | 6 | 3 | 0 | 0 | 0
Not completed — Subject/guardian decision | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase II Part
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted | Phase I: FGF401 80 mg + PDR001 300 mg | Phase I: FGF401 120 mg + PDR001 300 mg | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD | PhaseII: Group 3 - FGF401 120 mg QD
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 36 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 36 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 29 | 18
Not completed — Subject/guardian decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised all subjects who received at least one dose of study medication. Subjects enrolled in the Phase I part were analyzed according to the treatment they had been assigned to. Subjects enrolled in the Phase II part were analyzed by group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted | Phase I: FGF401 80 mg + PDR001 300 mg | Phase I: FGF401 120 mg + PDR001 300 mg | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD | PhaseII: Group 3 - FGF401 120 mg QD | Total
Number analyzed (Participants) | 11 | 6 | 5 | 26 | 19 | 7 | 6 | 6 | 30 | 36 | 20 | 172
Age, Customized [Number; unit: participants]
  18 y - <65 y | 6 | 4 | 3 | 14 | 12 | 4 | 3 | 3 | 22 | 15 | 10 | 96
  65 y - <85 y | 5 | 2 | 2 | 12 | 6 | 3 | 3 | 3 | 8 | 21 | 10 | 75
  >=85 y | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 3 | 6 | 0 | 1 | 4 | 8 | 7 | 12 | 47
  Male | 7 | 5 | 4 | 23 | 13 | 7 | 5 | 2 | 22 | 29 | 8 | 125
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 9 | 2 | 2 | 14 | 10 | 4 | 3 | 5 | 30 | 0 | 2 | 81
  Black | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Caucasian | 2 | 4 | 3 | 12 | 8 | 1 | 3 | 1 | 0 | 21 | 11 | 66
  Not applicable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 12 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT): Phase I Only
Description: A dose-limiting toxicity was defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurred within the evaluation period of DLTs and met any of the criteria listed. The estimation of the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of the treatment was based upon the estimation of the probability of DLT during the evaluation period for subjects in the dose determining set (DDS). A subject with multiple occurrences of a DLT under one treatment is counted only once in the AE category for that treatment. A subject with multiple DLTs within a primary system organ class is counted only once in the total row.
Time Frame: Cycle 1 (C1) (21 days) for FGF401 single agent, Cycle 1 and Cycle 2 (C2) (42 days) for FGF401 and PDR001 combination
Population: Dose Determining Set: All subjects from safety set (Phase I) who either met the minimum exposure criterion and had sufficient safety evaluations or had experienced a DLT during the DLT evaluation period.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted | Phase I: FGF401 80 mg + PDR001 300 mg | Phase I: FGF401 120 mg + PDR001 300 mg
Number analyzed (Participants) | 10 | 6 | 5 | 23 | 18 | 7 | 6 | 6
Percentage of participants
  Any Primary system organ class (SOC) | 10.0 | 0 | 0 | 4.3 | 5.6 | 42.9 | 0 | 0
  Invest.: Aspartate Aminotrans. increased | 0 | 0 | 0 | 4.3 | 0 | 42.9 | 0 | 0
  Invest.: Alanine aminotrans. increased | 10.0 | 0 | 0 | 0 | 0 | 14.3 | 0 | 0
  Invest.: Blood bilirubin increased | 0 | 0 | 0 | 0 | 5.6 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Phase I: 120 mg Fasted; Test type: Other; RP2D = 120 — The estimation parameter and recommended Phase 2 dose level for FGF401 (single agent - fasted) is 120mg
Statistical Analysis 2: Comparison: Phase I: 120 mg Fed; Test type: Other; RP2D = 120 — The estimation parameter and recommended Phase 2 dose level for FGF401 (single agent - fed) is 120mg
Statistical Analysis 3: Comparison: Phase I: FGF401 120 mg + PDR001 300 mg; Test type: Other; RP2D = 120 — The estimation parameter and recommended Phase 2 dose level for FGF401 + PDR001 combination is for FGF401 120mg
Statistical Analysis 4: Comparison: Phase I: FGF401 120 mg + PDR001 300 mg; Test type: Other; RP2D = 300 — The estimation parameter and recommended Phase 2 dose level for FGF401 + PDR001 combination is for PDR001 300mg

2. Primary Outcome: Time to Progression (TTP): Group 1 & Group 2 (Phase II Only)
Description: TTP is defined as the date of start treatment to the date of event defined as the first documented progression or death due to underlying cancer. Method used was Kaplan-Meier analysis.
  Group 1: HCC subjects form Asian countries; Group 2: HCC subjects form non-Asian countries
Time Frame: approx. 4.5 years
Population: Full Analysis Set (FAS): Comprised all subjects who received at least one dose of study medication. Subjects enrolled in the Phase II part were analyzed by group.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD
Number analyzed (Participants) | 30 | 36
months | 2.6 [1.3 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Interval for this Outcome Measure. Therefore, the upper limit is unavailable | 3.9 [2.9 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Intervals for this Outcome Measure. Therefore, the upper limit is unavailable

3. Primary Outcome: Overall Response Rate (ORR) Based on Local Assessment: Group 3 (Phase II Only)
Description: ORR is defined as the percentage of patients with a best overall response of CR or PR (RECIST v1.1).
  FGF401 single agent-Phase II part - Group 3 (non-HCC, other solid tumors).
Time Frame: approx. 4.5 years
Population: FAS: The full analysis set (FAS) comprised all subjects who received at least one dose of study medication. Subjects enrolled in the Phase II part were analyzed by group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PhaseII: Group 3 - FGF401 120 mg QD
Number analyzed (Participants) | 20
Percentage of participants | 0 [0.0 to 16.8]

4. Secondary Outcome: Best Overall Response (BOR) by Investigator Assessment: Phase I and Phase II
Description: BOR is the best response recorded from the start of the treatment until disease progression/recurrence. BOR is determined according to: complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD) and unknown.
Time Frame: approx. 4.5 years
Population: FAS: The full analysis set (FAS) comprised all subjects who received at least one dose of study medication. Subjects enrolled in the Phase I part were analyzed according to the treatment they had been assigned to. Subjects enrolled in the Phase II part were analyzed by group.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted | Phase I: FGF401 80 mg + PDR001 300 mg | Phase I: FGF401 120 mg + PDR001 300 mg | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD | PhaseII: Group 3 - FGF401 120 mg QD
Number analyzed (Participants) | 11 | 6 | 5 | 26 | 19 | 7 | 6 | 6 | 30 | 36 | 20
Participants
  Complete Response | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 0
  Stable Disease | 2 | 1 | 2 | 12 | 9 | 4 | 2 | 2 | 11 | 20 | 6
  Progressive Disease | 7 | 4 | 1 | 11 | 8 | 2 | 3 | 1 | 16 | 6 | 12
  Unknown | 2 | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 1 | 8 | 2

5. Secondary Outcome: Overall Response Rate (ORR) by Investigator Assessment Phase I and FGF401 Single Agent Phase II Groups 1 & 2
Description: ORR is defined as the proportion of patients with a best overall response of CR or PR (RECIST v1.1).
  Phase I part and FGF401 single agent Phase II Group 1 (HCC, Asians) and Group 2 (HCC, non-Asians)
Time Frame: approx. 4.5 years
Population: FAS: The FAS comprised all subjects who received at least one dose of study medication. Subjects enrolled in the Phase I part were analyzed according to the treatment they had been assigned to. Subjects enrolled in the Phase II part were analyzed by group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted | Phase I: FGF401 80 mg + PDR001 300 mg | Phase I: FGF401 120 mg + PDR001 300 mg | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD | PhaseII: Group 3 - FGF401 120 mg QD
Number analyzed (Participants) | 11 | 6 | 5 | 26 | 19 | 7 | 6 | 6 | 30 | 36 | 0
Percentage of participants | 0 [0.0 to 28.5] | 16.7 [0.4 to 64.1] | 20.0 [0.5 to 71.6] | 3.8 [0.1 to 19.6] | 0 [0.0 to 17.6] | 14.3 [0.4 to 57.9] | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 6.7 [0.8 to 22.1] | 5.6 [0.7 to 18.7] |

6. Secondary Outcome: Disease Control Rate (DCR) by Local Investigator Assessment Phase I and FGF401 Single Agent Phase II Groups 1, 2 & 3
Description: DCR is the percentage of participants with a best overall response of CR or PR or SD per local assessment according to RECIST v1.1. Phase I part and FGF401 single agent Phase II Group 1 (HCC, Asians) and Group 2 (HCC, non-Asians) and Group 3 (non-HCC, other solid tumors).
Time Frame: approx. 4.5 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted | Phase I: FGF401 80 mg + PDR001 300 mg | Phase I: FGF401 120 mg + PDR001 300 mg | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD | PhaseII: Group 3 - FGF401 120 mg QD
Number analyzed (Participants) | 11 | 6 | 5 | 26 | 19 | 7 | 6 | 6 | 30 | 36 | 20
percentage of participants | 18.2 [2.3 to 51.8] | 33.3 [4.3 to 77.7] | 60.0 [14.7 to 94.7] | 50.0 [29.9 to 70.1] | 47.4 [24.4 to 71.1] | 71.4 [29.0 to 96.3] | 50.0 [11.8 to 88.2] | 50.0 [11.8 to 88.2] | 43.3 [25.5 to 62.6] | 61.1 [43.5 to 76.9] | 30.0 [11.9 to 54.3]

7. Secondary Outcome: Time to Progression (TTP) in Participants Dosed With Single Agent FGF401 120 mg (Fasted & Fed) & With Combination FGF401 120 mg + PDR001 300 mg Q3W (Phase I)
Description: TTP is defined as the date of start treatment to the date of event defined as the first documented progression or death due to underlying cancer. Method used was Kaplan-Meier analysis.
Time Frame: approx. 4.5 years
Population: The full analysis set (FAS) comprised all subjects who received at least one dose of study medication. Subjects enrolled in the Phase I part were analyzed according to the treatment they had been assigned to.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: FGF401 120 mg + PDR001 300 mg
Number analyzed (Participants) | 26 | 19 | 6
months | 4.1 [1.6 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Interval for this Outcome Measure. Therefore, the upper limit is unavailable | 2.0 [1.4 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Interval for this Outcome Measure. Therefore, the upper limit is unavailable | 5.3 [3.0 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Interval for this Outcome Measure. Therefore, the upper limit is unavailable

8. Secondary Outcome: Overall Survival (OS) in Participants Dosed With Single Agent FGF401 120 mg (Fasted & Fed) and in Participants Dosed With Combination FGF401 120 mg and PDR001 300 mg Q3W (Phase I & II)
Description: Overall survival (OS) is defined as the time from date of start of treatment to date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last known date patient alive. Method used was Kaplan-Meier analysis.
Time Frame: start of treatment to death, up to about 53 months
Population: as for outcome 4
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: FGF401 120 mg + PDR001 300 mg | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD | PhaseII: Group 3 - FGF401 120 mg QD
Number analyzed (Participants) | 26 | 19 | 6 | 30 | 36 | 20
months | 7.0 [5.1 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Interval for this Outcome Measure. Therefore, the upper limit is unavailable | 4.9 [2.6 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Interval for this Outcome Measure. Therefore, the upper limit is unavailable | NA [NA to NA] — NA: did not observe enough events to calculate these parameters | 5.9 [5.1 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Interval for this Outcome Measure. Therefore, the upper limit is unavailable | 10.9 [7.9 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Interval for this Outcome Measure. Therefore, the upper limit is unavailable | 6.2 [4.2 to NA] — NA: it was pre-specified in the Statistical Plan to generate only one-sided 90% Confidence Interval for this Outcome Measure. Therefore, the upper limit is unavailable

9. Secondary Outcome: Progression-free Survival (PFS) - FGF401 Single Agent Phase II: Group 3
Description: Progression-free survival (PFS) is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient has not had an event, progression-free survival is censored at the date of last adequate tumor assessment. Group 3 - non-HCC, other solid tumors. Method used was Kaplan-Meier analysis.
Time Frame: 4.5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PhaseII: Group 3 - FGF401 120 mg QD
Number analyzed (Participants) | 20
months | 1.4 [1.4 to 2.8]

10. Secondary Outcome: Presence and/or Concentration of Anti-PDR001 Antibodies
Description: Serum PDR001 concentrations as well as immunogenicity analysis were performed for all subjects receiving PDR001. Treatment-induced ADA-positive percentage was based on percentage subjects ADA-negative at baseline. Treatment-boosted ADA-positive percentage was based on subjects ADA-positive at baseline.
Time Frame: Day 1 of Cycle 1 to 6, approx. 10 months after C1D1 and 150-day safety follow up (FU)
Population: FAS: The full analysis set (FAS) comprised all subjects who received at least one dose of study medication. Subjects enrolled in the Phase I part were analyzed according to the treatment they had been assigned to.
Measure: Number; unit: percentage of participants
Arm/Group | Phase II: Group 1 - FGF401 120 mg QD | Phase I: FGF401 120 mg + PDR001 300 mg
Number analyzed (Participants) | 6 | 6
percentage of participants
  ADA-negative | 100.0 | 83.3
  ADA-positive (i.e. ADA incidence) | 0 | 16.7
  Treatment-induced ADA-positive | 0 | 20.0
  Treatment-boosted ADA-positive | 0 | 0

11. Secondary Outcome: Cmax of PDR001 in Combination With FGF401: Phase I
Description: Cmax is the maximum (peak) observed plasma drug concentration (mass x volume-1)
Time Frame: After the first dosing sample collection was at: C1D1 0hr , C1D1 1hr, C1D8 168hr, C1D15 336hr, C2D1 504hr; each cycle is 21 days
Population: The PAS included all subjects who provided at least one evaluable drug concentration. For those requiring non-compartment analyses, the PAS included all subjects who provided an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Phase II: Group 1 - FGF401 120 mg QD | Phase I: FGF401 120 mg + PDR001 300 mg
Number analyzed (Participants) | 6 | 6
μg/mL | 74.7 (43.0) | 87.7 (5.4)

12. Secondary Outcome: AUClast and AUCtau of PDR001 in Combination of FGF401: Phase I
Description: AUClast: The AUC from time zero to the last measurable concentration sampling time (Tlast) (mass x time x volume-1)
  AUCtau (AUC0 504h): The AUC calculated to the end of a dosing interval (tau) (amount x time x volume-1)
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Phase II: Group 1 - FGF401 120 mg QD | Phase I: FGF401 120 mg + PDR001 300 mg
Number analyzed (Participants) | 6 | 6
day*μg/mL
  AUClast | 795 (34.5) | 978 (15.8)
  AUC0-504h (n = 3, 6): number analyzed (Participants) | 3 | 6
  AUC0-504h (n = 3, 6) | 760 (1.9) | 967 (13.9)

13. Secondary Outcome: T1/2 of PDR001: Phase I
Description: Due to the sparse PK sampling designed from PDR001, the PDR001 concentration data was insufficient for accurate estimation of secondary PK parameters including T1/2.
Time Frame: as for outcome 11
Population: The PAS incl. all subjects who provided at least one evaluable drug concentration. For those requiring non-compartment analyses, PAS incl. all subjects who provided an evaluable PK profile. Due to the sparse PK sampling designed for PDR001, PDR001 concentration data was insufficient for accurate estimation of secondary PK parameters including T1/2.
Arm/Group | Phase II: Group 1 - FGF401 120 mg QD | Phase I: FGF401 120 mg + PDR001 300 mg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Cmax of FGF401: Phase I
Description: Cmax is the maximum (peak) observed plasma drug concentration (mass x volume-1)
Time Frame: C1D1 (0 hour (h), 0.5h, 1h, 2h, 3h, 4h, 6h, 12h, 24h), C1D8 (0h, 0.5h, 1h, 2h, 3h, 4h, 6h, 12h, 24h), and C2D1 (0h, 0.5h, 1h, 2h, 3h, 4h, 6h, 12h, 24h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted
Number analyzed (Participants) | 10 | 6 | 5 | 26 | 19 | 7
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 6 | 5 | 5 | 26 | 19 | 7
  Cycle 1 Day 1 | 698 (36.1) | 967 (25.0) | 659 (15.2) | 1090 (37.9) | 1050 (32.3) | 1400 (32.1)
  Cycle 1 Day 8: number analyzed (Participants) | 7 | 6 | 4 | 24 | 18 | 6
  Cycle 1 Day 8 | 663 (46.8) | 838 (16.5) | 704 (22.1) | 1120 (36.5) | 1060 (22.1) | 1070 (46.0)
  Cycle 2 Day 1: number analyzed (Participants) | 9 | 6 | 5 | 22 | 17 | 4
  Cycle 2 Day 1 | 696 (44.2) | 786 (25.5) | 703 (41.7) | 1070 (32.2) | 1000 (23.9) | 1350 (28.1)

15. Secondary Outcome: Cmax of FGF401 in Combination With PDR001: Phase I
Description: Cmax is the maximum (peak) observed plasma drug concentration (mass x volume-1)
Time Frame: C1D1 (0h, 0.5h, 1h, 2h, 3h, 4h, 6h, 12h, 24h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase II: Group 1 - FGF401 120 mg QD | Phase I: FGF401 120 mg + PDR001 300 mg
Number analyzed (Participants) | 6 | 6
ng/mL | 732 (26.8) | 1450 (31.4)

16. Secondary Outcome: AUCinf, AUClast & AUCtau of FGF401: Phase I
Description: AUCinf: The AUC from time zero to infinity (mass x time x volume-1)
  AUClast: The AUC from time zero to the last measurable concentration sampling time (Tlast) (mass x time x volume-1)
  AUCtau: The AUC calculated to the end of a dosing interval (tau) (amount x time x volume-1)
Time Frame: C1D1 (0h, 0.5h, 1h, 2h, 3h, 4h, 6h, 12h, 24h), C1D8 (0h, 0.5h, 1h, 2h, 3h, 4h, 6h, 12h, 24h), and C2D1 (0h, 0.5h, 1h, 2h, 3h, 4h, 6h, 12h, 24h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted
Number analyzed (Participants) | 10 | 6 | 5 | 26 | 19 | 7
hr*ng/mL
  AUCinf C1D1: number analyzed (Participants) | 6 | 5 | 4 | 24 | 17 | 7
  AUCinf C1D1 | 4920 (51.9) | 5090 (32.9) | 5560 (23.1) | 7210 (35.4) | 8520 (35.2) | 8190 (42.7)
  AUClast C1D1: number analyzed (Participants) | 6 | 5 | 5 | 26 | 19 | 7
  AUClast C1D1 | 4610 (50.4) | 4710 (38.0) | 4600 (39.2) | 6710 (35.6) | 7850 (34.1) | 7920 (42.0)
  AUCtau C1D1: number analyzed (Participants) | 6 | 5 | 5 | 26 | 18 | 7
  AUCtau C1D1 | 4610 (50.4) | 4910 (30.3) | 4860 (29.4) | 6840 (33.6) | 8020 (33.5) | 7930 (41.8)
  AUCinf C1D8: number analyzed (Participants) | 6 | 6 | 4 | 18 | 15 | 6
  AUCinf C1D8 | 3650 (71.9) | 5130 (28.9) | 5550 (23.2) | 7590 (43.0) | 7980 (25.1) | 7850 (29.4)
  AUClast C1D8: number analyzed (Participants) | 6 | 6 | 4 | 24 | 18 | 6
  AUClast C1D8 | 3460 (62.5) | 4840 (27.0) | 5280 (23.9) | 6480 (47.5) | 7640 (33.1) | 7550 (28.6)
  AUCtau C1D8: number analyzed (Participants) | 7 | 6 | 4 | 24 | 16 | 6
  AUCtau C1D8 | 3650 (65.6) | 4850 (27.0) | 5290 (24.0) | 6970 (38.7) | 7330 (26.7) | 7510 (29.8)
  AUCinf C2D1: number analyzed (Participants) | 9 | 6 | 5 | 22 | 13 | 4
  AUCinf C2D1 | 4390 (54.0) | 4580 (30.6) | 5110 (44.3) | 7770 (33.2) | 8760 (23.5) | 7850 (25.7)
  AUClast C2D1: number analyzed (Participants) | 9 | 6 | 5 | 22 | 17 | 4
  AUClast C2D1 | 4100 (52.9) | 4210 (32.5) | 4880 (43.1) | 7260 (33.6) | 7520 (38.7) | 7610 (25.8)
  AUCtau C2D1: number analyzed (Participants) | 9 | 6 | 5 | 22 | 15 | 4
  AUCtau C2D1 | 4100 (52.7) | 4360 (28.5) | 4870 (43.7) | 7330 (31.7) | 7830 (23.4) | 7620 (25.7)

17. Secondary Outcome: AUCinf, AUClast & AUCtau of FGF401 in Combination With PDR001: Phase I
Description: as for outcome 16
Time Frame: C1D1 (0h, 0.5h, 1h, 2h, 3h, 4h, 6h, 12h, 24h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Phase II: Group 1 - FGF401 120 mg QD | Phase I: FGF401 120 mg + PDR001 300 mg
Number analyzed (Participants) | 6 | 6
hr*ng/mL
  AUCinf | 5030 (25.5) | 7540 (37.0)
  AUClast | 4760 (25.0) | 7280 (36.7)
  AUCtau | 4770 (24.4) | 7280 (36.7)

18. Secondary Outcome: T1/2 of FGF401: Phase I
Description: The elimination half-life associated with the terminal slope ( z) of a semi logarithmic concentration-time curve (time).
Time Frame: as for outcome 16
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (hr)
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted
Number analyzed (Participants) | 10 | 6 | 5 | 26 | 19 | 7
hour (hr)
  C1D1: number analyzed (Participants) | 6 | 5 | 4 | 24 | 17 | 7
  C1D1 | 6.27 (16.2) | 4.91 (31.6) | 5.2 (8.8) | 5.47 (14.4) | 5.16 (16.3) | 5 (11.3)
  C1D8: number analyzed (Participants) | 6 | 6 | 4 | 18 | 15 | 6
  C1D8 | 6.57 (16.6) | 6.08 (13.8) | 5.58 (12.0) | 5.43 (30.0) | 5.58 (17.1) | 5.24 (12.4)
  C2D1: number analyzed (Participants) | 9 | 6 | 5 | 22 | 13 | 4
  C2D1 | 6.46 (18.9) | 5.44 (34.9) | 5.43 (17.2) | 5.8 (22.1) | 5.81 (20.2) | 4.92 (14.4)

19. Post Hoc Outcome: All Collected Deaths
Description: This includes on-treatment deaths collected from first patient first treatment up to 30 days after drug discontinuation for a maximum of approx. 135.3 weeks (treatment duration ranged from 0.1 to 135.3 weeks for FGF401 single agent and from 6.0 to 57.0 weeks for FGF401 plus PDR001 combination). Deaths post treatment survival follow up were collected after the on treatment period, up to approx. 4.5 years. Participants who had not died after study drug discontinuation were censored at the last date when the participant had some documented personal contact (visit or phone call) with the investigator.
Time Frame: approx. 135.3 weeks, approx. 4.5 years
Population: as for outcome 3
Measure: Number; unit: Participants
Groups:
- All Patients of Single Agent FGF401: These were all the participants who received single dose of FGF401
- All Patients of Combination Dose: These were all the participants in the Phase I part who received combination dose of FGF401 and PDR001
- All Patients: Overall participants in the in Phase I & Phase II of study
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD | Phase II: Group 3 - FGF401 120 mg QD | All Patients of Single Agent FGF401 | Phase I: FGF401 80 mg + PDR001 300 mg | Phase I: FGF401 120 mg + PDR001 300 mg | All Patients of Combination Dose | All Patients
Number analyzed (Participants) | 11 | 6 | 5 | 26 | 19 | 7 | 30 | 36 | 20 | 160 | 6 | 6 | 12 | 172
Participants
  Total deaths | 10 | 5 | 3 | 23 | 12 | 4 | 20 | 22 | 16 | 115 | 2 | 2 | 4 | 119
  Deaths on-treatment | 2 | 1 | 0 | 4 | 6 | 1 | 2 | 2 | 2 | 20 | 0 | 0 | 0 | 20
  Deaths post-treatment survival follow up | 8 | 4 | 3 | 19 | 6 | 3 | 18 | 20 | 14 | 95 | 2 | 2 | 4 | 99

ADVERSE EVENTS:
Time Frame: This includes on-treatment deaths collected from first patient first treatment up to 30 days after drug discontinuation for a maximum of 135.3 weeks (treatment duration ranged from 0.1 to 135.3 weeks for FGF401 single agent and from 6.0 to 57.0 weeks for FGF401 plus PDR001 combination).
Description: Adverse Event (AE): Any sign or symptom that occurs during the study treatment plus the 30 or 150 days post treatment depending on single dose or combination dose.
Arm/Group | Phase I: 50 mg Fasted | Phase I: 80 mg Fasted | Phase I: 80 mg Fed | Phase I: 120 mg Fasted | Phase I: 120 mg Fed | Phase I: 150 mg Fasted | Phase II: Group 1 - FGF401 120 mg QD | Phase II: Group 2 - FGF401 120 mg QD | Phase II: Group 3 - FGF401 120 mg QD | All Patients of Single Agent FGF401 | Phase I: FGF401 80 mg + PDR001 300 mg | Phase I: FGF401 120 mg + PDR001 300 mg | All Patients of Combination Dose | All Patients
All-Cause Mortality (participants affected / at risk) | 2/11 | 1/6 | 0/5 | 4/26 | 6/19 | 1/7 | 2/30 | 2/36 | 2/20 | 20/160 | 0/6 | 0/6 | 0/12 | 20/172
Serious Adverse Events (participants affected / at risk) | 3/11 | 5/6 | 3/5 | 15/26 | 9/19 | 3/7 | 15/30 | 9/36 | 8/20 | 70/160 | 0/6 | 2/6 | 2/12 | 72/172
Other Adverse Events (participants affected / at risk) | 11/11 | 6/6 | 5/5 | 26/26 | 19/19 | 7/7 | 29/30 | 36/36 | 20/20 | 159/160 | 6/6 | 6/6 | 12/12 | 171/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: 50 mg Fasted (N=11) | Phase I: 80 mg Fasted (N=6) | Phase I: 80 mg Fed (N=5) | Phase I: 120 mg Fasted (N=26) | Phase I: 120 mg Fed (N=19) | Phase I: 150 mg Fasted (N=7) | Phase II: Group 1 - FGF401 120 mg QD (N=30) | Phase II: Group 2 - FGF401 120 mg QD (N=36) | Phase II: Group 3 - FGF401 120 mg QD (N=20) | All Patients of Single Agent FGF401 (N=160) | Phase I: FGF401 80 mg + PDR001 300 mg (N=6) | Phase I: FGF401 120 mg + PDR001 300 mg (N=6) | All Patients of Combination Dose (N=12) | All Patients (N=172)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 2 | 3 | 9 | 0 | 0 | 0 | 9
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Gastric varices (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 3
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 2 | 2 | 5
Biloma (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hepatic haematoma (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Inferior vena caval occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: 50 mg Fasted (N=11) | Phase I: 80 mg Fasted (N=6) | Phase I: 80 mg Fed (N=5) | Phase I: 120 mg Fasted (N=26) | Phase I: 120 mg Fed (N=19) | Phase I: 150 mg Fasted (N=7) | Phase II: Group 1 - FGF401 120 mg QD (N=30) | Phase II: Group 2 - FGF401 120 mg QD (N=36) | Phase II: Group 3 - FGF401 120 mg QD (N=20) | All Patients of Single Agent FGF401 (N=160) | Phase I: FGF401 80 mg + PDR001 300 mg (N=6) | Phase I: FGF401 120 mg + PDR001 300 mg (N=6) | All Patients of Combination Dose (N=12) | All Patients (N=172)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 2 | 1 | 5 | 1 | 5 | 18 | 2 | 2 | 4 | 22
Hyperglobulinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 0 | 3 | 3 | 1 | 1 | 13 | 0 | 3 | 3 | 16
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 4 | 0 | 5 | 6 | 9 | 31 | 0 | 2 | 2 | 33
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 7 | 1 | 0 | 5 | 5 | 1 | 21 | 0 | 0 | 0 | 21
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 2 | 5 | 0 | 2 | 4 | 3 | 2 | 19 | 0 | 0 | 0 | 19
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 1 | 0 | 5 | 5 | 6 | 23 | 1 | 0 | 1 | 24
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 4 | 18 | 14 | 7 | 23 | 23 | 17 | 118 | 3 | 4 | 7 | 125
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 5 | 0 | 0 | 0 | 5
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4 | 0 | 0 | 0 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 5 | 0 | 0 | 0 | 5
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 6 | 0 | 0 | 0 | 6
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 5 | 6 | 1 | 7 | 6 | 11 | 38 | 0 | 2 | 2 | 40
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 4
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 6 | 1 | 5 | 4 | 9 | 32 | 0 | 1 | 1 | 33
Asthenia (General disorders) | 2 | 2 | 0 | 4 | 3 | 2 | 3 | 6 | 4 | 26 | 0 | 0 | 0 | 26
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 5 | 0 | 0 | 0 | 5
Fatigue (General disorders) | 2 | 1 | 0 | 6 | 4 | 0 | 2 | 8 | 7 | 30 | 1 | 2 | 3 | 33
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2
Hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 3
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 3
Oedema peripheral (General disorders) | 0 | 1 | 0 | 9 | 0 | 0 | 8 | 9 | 3 | 30 | 0 | 2 | 2 | 32
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 4 | 0 | 0 | 0 | 4
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 3 | 0 | 2 | 6 | 1 | 1 | 9 | 4 | 5 | 31 | 1 | 3 | 4 | 35
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 5 | 0 | 0 | 0 | 5
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 3
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 3
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 3
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 3
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 5 | 2 | 0 | 2 | 7
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 4 | 0 | 0 | 0 | 4
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 5 | 0 | 0 | 0 | 5
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 0 | 0 | 4
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 1 | 7 | 0 | 0 | 0 | 7
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 3 | 3 | 2 | 14 | 11 | 7 | 13 | 11 | 6 | 70 | 0 | 4 | 4 | 74
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4 | 0 | 0 | 0 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 2 | 16 | 14 | 7 | 14 | 11 | 5 | 76 | 1 | 5 | 6 | 82
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 4 | 5 | 1 | 4 | 2 | 2 | 20 | 0 | 1 | 1 | 21
Blood bilirubin increased (Investigations) | 4 | 3 | 1 | 11 | 2 | 0 | 6 | 3 | 1 | 31 | 1 | 2 | 3 | 34
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 5 | 0 | 1 | 1 | 6
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 1 | 5
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 4 | 2 | 0 | 4 | 3 | 3 | 17 | 1 | 1 | 2 | 19
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 4 | 6 | 1 | 14 | 0 | 0 | 0 | 14
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 2 | 4
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 6 | 0 | 1 | 1 | 7
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 3
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 4 | 4 | 12 | 0 | 1 | 1 | 13
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 0 | 10 | 2 | 4 | 6 | 9 | 12 | 47 | 0 | 0 | 0 | 47
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 5 | 0 | 0 | 0 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 3
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 6 | 0 | 0 | 0 | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 8 | 2 | 3 | 5 | 13
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 7 | 1 | 2 | 14 | 0 | 0 | 0 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 5 | 0 | 1 | 1 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 7 | 1 | 0 | 1 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 3
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 1 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 5 | 4 | 1 | 14 | 2 | 0 | 2 | 16
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 1 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 3 | 2 | 3 | 12 | 0 | 0 | 0 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 4 | 0 | 1 | 1 | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 3
Dysgeusia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 6 | 0 | 1 | 1 | 7
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 3 | 3 | 12 | 0 | 1 | 1 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 5 | 0 | 0 | 0 | 5
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 4 | 2 | 5 | 16 | 0 | 1 | 1 | 17
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Varicocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 2 | 2 | 7 | 3 | 2 | 19 | 0 | 1 | 1 | 20
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | 0 | 1 | 4 | 3 | 3 | 17 | 0 | 0 | 0 | 17
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 5 | 0 | 0 | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 4 | 0 | 0 | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 6 | 0 | 1 | 1 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 2 | 7 | 1 | 0 | 1 | 8
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 4 | 5 | 1 | 5 | 8 | 0 | 28 | 0 | 2 | 2 | 30
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 6 | 0 | 2 | 2 | 8
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3 | 2 | 9 | 0 | 0 | 0 | 9
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT02325739/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT02325739/SAP_001.pdf